CLINICAL TRIAL: NCT05989178
Title: Prospective Recurrent Pregnancy Loss (ProRPL) Registry
Brief Title: Prospective Recurrent Pregnancy Loss Registry
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mohamed Bedaiwy, Principal Investigator, Professor and Head Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynaecology, University of British Columbia, University of British Columbia
Other Study IDs: H21-01887
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Recurrent pregnancy loss; Unexplained; Explained; Miscarriage; Live Birth
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Routinely Collected Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Products of conception (optional)
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: Data Registry — Follow-up questionnaires sent every year for the 5 years following the patient's initial visit.

SUMMARY:
The purpose of this Registry is to prospectively collect data of Recurrent Pregnancy Loss (RPL) patients attending the specialized care centre at the BC Women's Hospital, in order to evaluate investigation practices, treatment options, and outcomes for this patient population over time.

DETAILED DESCRIPTION:
The Recurrent Pregnancy Loss Program at the BC Women's Centre for Reproductive Health is the only tertiary care centre of its kind in British Columbia, and has provided specialized and comprehensive care to RPL patients for the past 15 years. Using a team-based collaborative model, the program provides point-of-care investigations, surgical treatment, clinical management, education, and grief counselling.

All RPL patients are asked to complete the intake questionnaire prior to their initial visit at the clinic. If the patient provides their consent to take part in research, their data will be copied from the clinical database to the research database. The questionnaire includes information regarding patient demographics, obstetric history, gynecological history, personal and medical history, family history and partner information. Additionally, data will also be collected from patient charts, follow-up questionnaires sent once a year for the next 5 years following the patient's initial visit, and medical records from fertility clinics and general practitioners when available.

The online data registry is housed in the Research Electronic Data Capture (REDCap) platform located at BC Children's Hospital (BCCH).

As an optional component of this study, patients invited to join the registry will also be presented with the option to register with the BCCH BioBank to store their tissue samples collected in the RPL clinic for clinical & diagnostic purposes.

ELIGIBILITY:
Inclusion Criteria:

• Patients seen at the BC Women's Recurrent Pregnancy Loss Clinic with recurrent pregnancy loss, defined as ≥2 pregnancy losses before 20 weeks of gestation.

Exclusion Criteria:

• Patients at BC Women's Recurrent Pregnancy Loss Clinic seen for reasons other than recurrent pregnancy loss.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients at the BC Women's Recurrent Pregnancy Loss Clinic seen for recurrent pregnancy loss.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Live Birth | 5 years
  Percent of patients with a live birth within 5 years after initial visit at the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Bedaiwy, MD, PhD, Principal Investigator — BC Women's Hospital & Health Centre
Locations (1):
- BC Women's Hospital & Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No